CLINICAL TRIAL: NCT04129905
Title: Assessment of the Relations Between Endothelial and Venous Dysfunctions and Left Ventricular Obstruction in Genetic Hypertrophic Cardiomyopathies
Acronym: HCM-Vein
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Fédération Française de Cardiologie (Other); Fondation Bordeaux Université (Unknown); Amicus Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CHUBX 2018/04
Record Dates: First submitted 2019-06-12; First posted 2019-10-17 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: Hypertrophic Cardiomyopathy; Endothelial Dysfunction
Keywords: Hypertrophic Cardiomyopathy; Endothelial Dysfunction; Venous return; Left ventricular outflow-tract obstruction; Sudden cardiac death risk
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic; Ventricular Outflow Obstruction, Left | interventions — Electrocardiography; Electrocardiography, Ambulatory; Echocardiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Symptomatic HCM patients (Experimental): 30 subjects (25-26 sarcomeric, 4-5 Fabry).
  Interventions: Biological: BNP blood sample test; Diagnostic Test: Electrocardiogram; Diagnostic Test: Holter ECG; Diagnostic Test: Echocardiography; Diagnostic Test: Air venous plethysmography; Diagnostic Test: Upper member arterial Doppler echography with analysis of FMD; Biological: Endothelial function biomarkers
- Healthy controls subjects (Active Comparator): 10 subjects (matched in age and sex to HCM patients) to obtain reference values of endothelial dysfunction.
  Interventions: Diagnostic Test: Air venous plethysmography; Diagnostic Test: Upper member arterial Doppler echography with analysis of FMD; Biological: Endothelial function biomarkers

INTERVENTIONS:
Biological: BNP blood sample test — Performed during normal recommended follow-up of the HCM patients.
  Arms: Symptomatic HCM patients
Diagnostic Test: Electrocardiogram — Performed during normal recommended follow-up of the HCM patients.
  Arms: Symptomatic HCM patients
Diagnostic Test: Holter ECG — Performed during normal recommended follow-up of the HCM patients.
  Arms: Symptomatic HCM patients
Diagnostic Test: Echocardiography — Performed during normal recommended follow-up of the HCM patients. Echocardiography at rest and during exercise.
  Arms: Symptomatic HCM patients
Diagnostic Test: Air venous plethysmography — Performed specifically for the research. Non invasive, and non painful test evaluating different parameters of venous filling by inflation of an armband around the leg, upright positioning, flexion-extension of the leg. Total duration estimated at 30-45 minute.
Diagnostic Test: Upper member arterial Doppler echography with analysis of FMD — Performed specifically for the research. Measurement of the evolution of brachial artery diameter before and after inflation of a armband during 5 minutes. Non invasive and non painful test, duration 30 minutes.
Biological: Endothelial function biomarkers — Performed specifically for the research. Blood sample test, 5 minutes.

SUMMARY:
Left ventricular obstruction is an invalidating complication of hypertrophic cardiomyopathies (HCM), and endothelial dysfunction has also been observed in these pathologies. However, the relation between obstruction and endothelial and venous dysfunctions has not been previously studied.

The main objective is to investigate the relations between endothelial and venous dysfunctions and symptomatic left ventricular outflow-tract obstruction in HCM patients.

DETAILED DESCRIPTION:
Hypertrophic cardiomyopathies (HCM) secondary to sarcomeric gene mutation or to Anderson-Fabry disease can be complicated by left ventricular (LV) outflow-tract obstruction responsible of disabling exercise symptoms. LV outflow-tract obstruction is a complex, multifactorial and dynamical phenomenon influenced by the degree of LV hypertrophy but also by mitral valve elongation and hemodynamical components including venous return (LV preload). The clinical and research team of Dr Réant, responsible of the Bordeaux Competence Center in hereditary or rare Cardiomyopathies, has recently demonstrated that LV outflow-tract obstruction can also be influenced by the conditions of realization of exercise echocardiography tests (position: upright versus supine, type: bicycle versus treadmill), and by an abnormal venous return capacity. In parallel, it has also been demonstrated, by other research teams, that HCM can be associated to endothelial and microvascular peripheral dysfunctions. However, to date, the relation between these two elements, and with sudden cardiac death risk, have not been previously studied.

The tests which will be performed during normal recommended follow-up of the HCM patients will be: Brain Natriuretic Peptide (BNP) blood sample test, electrocardiogram (ECG), Holter ECG, echocardiography at rest and during exercise.

The tests realized in addition will be:

* air venous plethysmography: non invasive, and non painful test evaluating different parameters of venous filling by inflation of an armband around the leg, upright positioning, flexion-extension of the leg. Total duration estimated at 30-45 minutes.
* upper member arterial Doppler echography with analysis of Flow Mediated Dilatation (FMD) : measurement of the evolution of brachial artery diameter before and after inflation of a armband during 5 minutes. Non invasive and non painful test, duration 30 minutes..
* endothelial function biomarkers: blood sample test, 5 minutes. No follow-up is required for this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients and volunteers:

  * Adults (age ≥18 years), male or female,
  * For female in age, efficient contraception will be required and a negative pregnancy test will be required,
  * Signed informed consent form will required for each included subject after having read the information note,
  * Affiliated to the national social security system,
* Patients:

  .Patients diagnosed to have HCM secondary to sarcomeric mutation or to Fabry disease, symptomatic (dyspnea on exertion and/or chest pains during exercise),
* Healthy volunteers:

  * Subjects without known cardiac disease,
  * No smokers.

Exclusion Criteria:

* Patients and volunteers:

  * No cardiac pathology reducing life expectancy to less than 12 months (cancer),
  * Unbalanced arterial hypertension (systolic >160 mmHg and/or diastolic >120 mmHg),
  * Pregnancy or breastfeeding,
  * Major obesity > 140 kg,
  * Impossibility or refusal to give or sign the consent form,
  * Subject in period of exclusion relative to an other protocol,
  * Subject deprived of liberty by judicial or administrative decision,
  * Major protected by the Law
* Patients:

  * Atrial fibrillation at the time of inclusion
  * Valvulopathy with severity greater than moderate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-10-22 (Actual); Primary Completion 2021-12-14 (Actual); Study Completion 2021-12-14 (Actual)

PRIMARY OUTCOMES:
Assessment of the venous ejection fraction | Day 0
  Via a plethysmography exam. The venous ejection fraction is measured in percentage.
Assessment of the caliber variation of the brachial artery | Day 0
  Via a recording of arterial Doppler echography with analysis of FMD parameters. This parameter is measured in percentage.
Measure of the Willebrand factor | Day 0
  The analysis of this biomarker of endothelial function is performed via a peripheral venous sample.
  This biomarker is measured in percentage.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia REANT, MD, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- University Hospital, Bordeaux, Pessac, France